CLINICAL TRIAL: NCT05153213
Title: Correlation of Length of Index Finger to Vertical Dimensions of Occlusion for Edentulous Patients and Assessment of Patient Satisfaction - A Randomized Clinical Trial
Brief Title: Correlation of Length of Index Finger to Vertical Dimensions of Occlusion for Edentulous Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shujah Adil Khan, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKhanDowUHS
Record Dates: First submitted 2021-03-23; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Patient Satisfaction; Dental Prosthesis; Edentulous Jaw
Keywords: Occlusal vertical dimension, edentulous patients,
MeSH Terms: conditions — Patient Satisfaction; Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finger Lengths (Experimental): Vernier caliper was used to determine the length of Index Finger to record Vertical Dimensions of Occlusion
  Interventions: Procedure: Finger lengths
- Conventional method (Active Comparator): Willis gauge was used to determine the Length from Base of the nose to Base of the chin to record Vertical Dimensions of Occlusion
  Interventions: Procedure: Conventional method

INTERVENTIONS:
Procedure: Finger lengths — Vernier caliper was used to measure finger length
  Arms: Finger Lengths
Procedure: Conventional method — Gillis gauge was used to measure occlusal vertical dimension
  Arms: Conventional method

SUMMARY:
This study is a randomized clinical trial comparing the conventional method of recording occlusal vertical dimension using Willis gauge from the base of the nose to the base of the chin with the other method using vernier caliper for the length of the index finger to access the satisfaction level of edentulous patients acquiring complete dentures.

DETAILED DESCRIPTION:
This study was to apply the anthropometric methods to correlate the length of fingers to occlusal vertical dimensions and also by using the Willis Method to assess the occlusal vertical dimension for edentulous patients and assess satisfaction by comparing both the methods for patients who are in the process of acquiring complete dentures. Furthermore, conventional methods are applied most commonly for the recording of occlusal vertical dimensions. This study also bridged the knowledge gap among clinicians to adapt to a different methodology for recording the VDO using the anthropometric measurement of fingers which would improve denture satisfaction. Therefore, a total of 71 patients were selected for this study, having lost their OVD due to the complete absence of teeth and having no history of maxillofacial or orthognathic surgery, nor any skeletal deformities or disfigurement of fingers. The measurements were made at the appointment for jaw relations records in which the length of the fingers was measured with a digital Vernier caliper and also the conventional methods were applied for recording the occluding vertical dimensions which included recording the distance from the base of the nose septum (Subnasion - Sn) to the base of the chin (Menton - Me) (Sn-Me). The length of the index finger (2D) was recorded and a correlation was found between Sn-Me and finger length.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients
* Patients willing to participate in the study
* Male patients without a beard

Exclusion Criteria:

* Partially dentate patients
* Patients having any maxillofacial or myofascial disorders
* Any history of orthognathic or orthodontic surgery
* Deformities or disfigurement of fingers
* Patients with neurological problems in the head and neck
* Any bony defects or visible sharp spicules
* Nose or chin deformity
* TMJ disorders (intracapsular/extracapsular)
* Heavy bulky chin area (double chin)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Complete Dentures | 6 Months
  Satisfaction with Complete Dentures after assessment of occlusal vertical dimension with Length of Index Finger

CONTACTS AND LOCATIONS:
Overall Officials: Shujah A Khan, BDS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhajj MN, Khalifa N, Abduo J, Amran AG, Ismail IA. Determination of occlusal vertical dimension for complete dentures patients: an updated review. J Oral Rehabil. 2017 Nov;44(11):896-907. doi: 10.1111/joor.12522. Epub 2017 Jun 10. PMID 28600914
- [Derived] Khan SA, Raza Kazmi SM, Ahmed S, Hani U, Choudhry Z, Sukkurwala A. Correlation of index finger length to vertical dimensions of occlusion for edentulous patients and their satisfaction: a randomized controlled trial. Sci Rep. 2023 May 7;13(1):7414. doi: 10.1038/s41598-023-33722-x. PMID 37150797